CLINICAL TRIAL: NCT06748807
Title: Physiological Effects of Early Pathophysiology-driven Airway Pressure Release Ventilation (APRVplus) and Time-Controlled Adaptive Ventilation (TCAV) in Acute Respiratory Distress Syndrome (ARDS): a Randomized Crossover Clinical Trial
Brief Title: Physiological Effects of APRVplus and TCAV in ARDS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: West China Hospital (Other)
Responsible Party: Principal Investigator, Zhou Yongfang, Zhou Yongfang, Sichuan University
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Supportive Care
Other Study IDs: 2023 approved No.193
Record Dates: First submitted 2024-12-19; First posted 2024-12-27 (Actual); Last update posted 2024-12-27 (Actual); Status verified 2024-12

CONDITIONS: ARDS (Acute Respiratory Distress Syndrome)
MeSH Terms: conditions — Acute Lung Injury

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- APRVplus (Experimental): An Early Pathophysiology-driven Airway Pressure Release Ventilation
  Interventions: Procedure: APRVplus
- TCAV (Other): Time Controlled Adaptive Ventilation (TCAV)
  Interventions: Procedure: TCAV

INTERVENTIONS:
Procedure: APRVplus — Early Pathophysiology-driven Airway Pressure Release Ventilation (APRVplus)
  Arms: APRVplus
Procedure: TCAV — Time-Controlled Adaptive Ventilation (TCAV)
  Arms: TCAV

SUMMARY:
In previous studies, airway pressure release ventilation (APRV) has been proven to be an important respiratory support method for ARDS patients, and various APRV ventilation strategies have been proposed. This study aims to compare the physiological effects of two types of APRV ventilation strategy, Early Pathophysiology-driven APRV (APRVplus) and Time-Controlled Adaptive Ventilation (TCAV), through randomized crossover trials, providing evidence for clinical application and further research on APRV.

ELIGIBILITY:
Inclusion Criteria:

* intubated and mechanically ventilated patients
* meet the 2023 global new definition of ARDS

Exclusion Criteria:

* Pregnancy
* The expected duration of mechanical ventilation was less than 48 hours
* Intracranial hypertension (suspected or confirmed)
* Neuromuscular disorders that are known to prolong the need for mechanical ventilation
* Known or suspected chronic obstructive pulmonary disease(COPD)
* Terminal stage of disease
* Pneumothorax (drained or not)at enrollment
* Treatment with extracorporeal support (ECMO) at enrollment
* There was a lack of commitment to life support

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2023-12-15 (Actual); Primary Completion 2024-12-15 (Actual); Study Completion 2024-12-15 (Actual)

PRIMARY OUTCOMES:
△PL（PLThigh - PLTlow) | during the mechanical ventilation procedure
  Transpulmonary pressure swings (△PL) equal to PLThigh - PLTlow

SECONDARY OUTCOMES:
EtCO2 | during the mechanical ventilation procedure
  end-tidal carbon dioxide
GI | during the mechanical ventilation procedure
  global inhomogeneity
PaO2(mmHg) | during the mechanical ventilation procedure
  the arterial partial pressure of oxygen

CONTACTS AND LOCATIONS:
Locations (1):
- West China Hospital, Sichuan University, Chengdu, Sichuan, China

IPD SHARING:
Plan to Share IPD: Undecided